CLINICAL TRIAL: NCT03553979
Title: Project Grip&Health: A Behavioural Intervention Which Uses an Integral Approach to Reduce Stress, Smoking, Improve Financial Health and Self-perceived Health of Low SES-residents in Rotterdam
Brief Title: Grip&Health: Behavioural Intervention to Reduce Smoking, Stress and Improve Financial Health in Low-SES in Rotterdam
Acronym: Grip&Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Indigo Rijnmond, the Netherlands (Unknown); Avant Sanare, The Netherlands (Unknown); Erasmus University Rotterdam (Other)
Responsible Party: Principal Investigator, Ingmar Franken, Professor, Erasmus Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: FNO projectnr. 102291
Record Dates: First submitted 2018-01-08; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Smoking Cessation; Smoking, Cigarette; Smoking; Stress; Stress, Psychological; Health Behavior; Smoking, Tobacco
Keywords: stress management; stress intervention; smoking intervention; lower SES; lower income
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking; Smoking; Stress, Psychological; Health Behavior; Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: Stress management program (SM) Stress management and Buddy program (SM-B)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stress management program (SM) (Experimental): The stress management program (SM) is a program which has been tailored to meet the specific needs of low-SES participants. The SM consists of 4-weekly sessions (1.5hours/session) and a follow-up session 8 weeks later. A core element of SM is its group-based format in which psycho-educative topics on stress responses and coping and motivation to stop smoking link up with cognitive and behavioural technique activities.
  Interventions: Behavioral: Stress management program (SM)
- Stress management + Buddy program (SM-B) (Experimental): The stress management + buddy program (SM-B) includes the same psycho-educative topics and exercises, cognitive and behavioural technique activities as the SM condition. The SM-B in addition to SM utilises one-to-one support through a buddy selected by a participant. A buddy, 18 year or older is a student or a volunteer who is recruited and trained by Indigo Rijnmond. The buddy pairs up with a participant and provides the following: supports participant in managing and filling in tax/welfare papers; 2) helps a participant to get a grip over his/her personal finances; and 3) helps a participant to overcome daily barriers (eg. arranging childcare). Over the duration of the course, the buddy meets up 6 times with a participant every second week in a public area.
  Interventions: Behavioral: Stress management + Buddy program (SM-B)
- Control (No Intervention): Participants in the control condition are instructed to continue with their normal daily behaviour. They will be invited to complete the questionnaires and objective measurements at the equivalent times as the intervention groups, thus at baseline, 4 weeks after baseline and 12 weeks after baseline. After the control period, participants in the control condition will be offered the intervention.

INTERVENTIONS:
Behavioral: Stress management program (SM) — Participants follow the SM program.
  Arms: Stress management program (SM)
Behavioral: Stress management + Buddy program (SM-B) — In addition to receiving the SM, participants in the SM-B will also receive one-to-one support through a buddy.
  Arms: Stress management + Buddy program (SM-B)

SUMMARY:
Grip&Health: randomised trial which will examine the effect of theory-based multicomponent behavioural intervention for reducing stress, smoking and improving financial health and perceived health of low-SES residents in Rotterdam. Between January 2018 and July 2018, a total of 300 participants will be recruited and randomised either to a stress management program (SM), stress management with a buddy program (SM-B) or a control condition. The investigators hypothesise that compared to participants in the control condition, participants in the intervention arms will demonstrate reduced stress, reduced smoking and improved financial health and perceived health.

ELIGIBILITY:
Inclusion Criteria:

* perceive stress
* smoke
* poor financial health

Exclusion Criteria:

* follow other stress management course
* follow smoking cessation course
* receive help from debt services for their financial problems
* have health problems which hamper their ability to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported Stress | at baseline (T0), 4 weeks after baseline (T1) and 12 weeks after baseline (T2)
  Change in self-reported Stress.
  The Depression, Anxiety and Stress (DASS) questionnaire will be used to measure change in self-reported stress from baseline (T0), at 4 weeks after baseline (T1) and at 12 weeks after baseline (T2).
  The DASS is a 21-item questionnaire with three self-report scales (Depression, Anxiety and Stress). Scores for depression, anxiety and stress are determined by summing the scores of the 21 items. Ranges for depression, anxiety and stress are 0-28, 0-20, and 0-33, respectively. Lower scores indicate less severity.
  In this study participants will be asked to complete the DASS-21 questionnaire at three different time points (T0, T1 and T2). This is done so the investigators can assess the change in scores of self-reported stress across time points (T0, T1 and T2).
Objective Stress | at baseline (T0), 4 weeks after baseline (T1) and 12 weeks after baseline (T2)
  Change in objective evaluations of stress based on heart rate variability (HRV) from baseline (T0), at 4 weeks after baseline (T1) and at 12 weeks after baseline (T2).
  HRV indicates variability of time intervals between two consecutive heartbeats with each heartbeat having a R-wave which peaks in the R peak. The variations between two RR intervals are defined as HRV. A higher HRV value reflects a greater variation of the RR whereas a lower HRV indicates small variation.
  Participants beat-to-beat heart rate is measured using wrist wearables provided by Philips. During the measurements, the wearables are mounted on a participant's wrist and the participant is instructed to sit in a resting state for five minutes while the beat-to-beat heart rate is recorded. HRV analysis is derived from the recorded data using an appropriate software program. To assess change over time points (T0, T1 and T2), participants's beat-to-beat heart rate will be measured at three time points
Self-reported Smoking | at baseline (T0), 4 weeks after baseline (T1) and 12 weeks after baseline (T2)
  Change in self-reported Smoking.
  The Global Adult Tobacco Survey (GATS) questionnaire will be used to measure change in self-reported smoking from baseline (T0), at 4 weeks after baseline (T1) and at 12 weeks after baseline (T2).
  Participants will be asked to complete the questionnaire at three time points (T0, T1 and T2). This is done so the investigators can assess the change in self-reported smoking across time points.
Dependence of nicotine | at baseline (T0), 4 weeks after baseline (T1) and 12 weeks after baseline (T2)
  Fagerstrom Test for Nicotine Dependence (FTND) questionnaire will be used to measure change in level of nicotine dependence from baseline (T0), at 4 weeks after baseline (T1) and at 12 weeks after baseline (T2).
  The FTND test is used to assess the intensity of physical addiction to nicotine. The test is designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. It contains six items that evaluates the quantity of cigarette consumption, the compulsion to use and dependence. Yes/No items on FTND are scores from 0-1 and multiple choice items are scores from 0-3. The items are summed to yield a total score of 0-10. The higher the FTND, the more intense a participant's physical dependence on nicotine.
  In this study, participants will be asked to complete the FTND at three time points (T0, T1 and T2). This is done so the investigators can assess the change in the level of nicotine dependence across time points.
Carbon Monoxide breath test | at baseline (T0), 4 weeks after baseline (T1) and 12 weeks after baseline (T2)
  Change in exhaled Carbon Monoxide (CO) levels from baseline (T0), at 4 weeks after baseline (T1) and at 12 weeks after baseline (T2).
  The CO breath test is a biological method used to verify smoking or non-smoking status of participants.
  In this study, participants's exhaled CO levels will be measured (Micro SmokeLyzer; Bedfont, UK). A CO level ≥10 ppm reflects a heavy smoker. During the measurements, participants are instructed to hold their breath for 15 seconds and subsequently to slowly exhale into a mouthpiece connected to the SmokeLyzer device until their lungs are empty.
  Participants CO levels will be recorded at three time points (T0, T1 and T2). This is done so the investigators can assess the change in C0 levels across time points.
Self-perceived health | at baseline (T0), 4 weeks after baseline (T1) and 12 weeks after baseline (T2)
  The Short Form Health Survey version 2 (SF-12v2) questionnaire will be used to measure change in self-perceived health from baseline (T0), at 4 weeks after baseline (T1) and at 12 weeks after baseline (T2).
  The SF-12v2 is a 12-item with three dimensions both for functioning (physical, social and role) and for wellbeing (mental health, general health perceptions and pain). In this study, participants will be asked to rate their general health on a Likert-type scale (1=poor, 2=fair, 3= good, 4= very good, and 5=excellent). Low scores (poor) on the general health scale represent a person who believes his/her health to be poor and high score (excellent) represents someone who sees his/her health as excellent.
  Participants will be asked to complete the SF-12v2 questionnaire at three time points (T0, T1 and T2). This is done so the investigators can assess the change in health perceptions across time points.
Financial health | at baseline (T0), 4 weeks after baseline (T1) and 12 weeks after baseline (T2)
  Change in participant's's financial health will be measured from baseline (T0), at 4 weeks after baseline (T1) and at 12 weeks after baseline (T2).
  In this study, participants's financial health will be measured by asking them to report: 1) their total monthly income; 2) their spouse/partner's total monthly income; and 3) money shortages experienced in the past month.
  Participants will be asked to fill this questionnaire in at three time points (T0, T1 and T2). This is done to assess changes in financial health across time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University College, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Shagiwal SS, Schop-Etman A, Bergwerff I, Vrencken W, Denktas S. The BeHealthyR Study: a randomized trial of a multicomponent intervention to reduce stress, smoking and improve financial health of low-income residents in Rotterdam. BMC Public Health. 2018 Jul 18;18(1):891. doi: 10.1186/s12889-018-5728-7. PMID 30021551